CLINICAL TRIAL: NCT03304574
Title: CheckED Yourself: Using Emergency Department Screening to Impact Adolescent Risk Behavior
Brief Title: CheckED Yourself Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Taraneh Shafii, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00000365
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Adolescent Behavior; Risk Behavior; Motivation
MeSH Terms: conditions — Adolescent Behavior; Risk-Taking

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups, a control or intervention group. Those assigned to the control group will complete the electronic health assessment only and will not receive integrated personalized feedback. Those assigned to the intervention group will complete the electronic health assessment and will receive integrated personalized feedback.
Who Masked: Participant
Masking Description: Participants will be blinded to their group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will complete the electronic health assessment only and will not receive integrated personalized feedback
- Intervention (Experimental): Participants will complete the electronic health assessment and will receive integrated personalized feedback
  Interventions: Behavioral: Integrated personalized feedback

INTERVENTIONS:
Behavioral: Integrated personalized feedback — Integrated personalized feedback about self-reported risk behaviors will be generated and shown to participants as they complete their baseline health risk assessment using the CheckED Yourself app. The integrated personalized feedback is based on motivational feedback strategies such as normative feedback (comparison to peer behaviors and age-based health guidelines), increasing knowledge regarding potential consequences of behaviors, and providing practical tips for changing behavior.
  Arms: Intervention

SUMMARY:
During adolescence, the most common causes of morbidity and mortality are related to risky behaviors. The American Academy of Pediatrics recommends that adolescents be screened for these behaviors during primary care visits, but many adolescents do not receive the recommended risk behavior screening and counseling, in part because they are infrequently seen in primary care. The objective of this study is to evaluate if the electronic health screening tool, which includes an electronic health assessment with integrated personalized feedback, reduces risk behaviors in adolescents seen in the Emergency Department (ED).

DETAILED DESCRIPTION:
Adolescents and their parents (if participant is under the age of 18 years) will be approached and invited to participate in the study during their Emergency Department (ED) visit. Following consent, adolescents will be randomized to the intervention or control group. A tablet computer will be provided to the participants for use during their baseline assessment in the ED. The CheckED Yourself App will be pre-loaded on the tablet. The CheckED Yourself App (eHA-IPF) is an innovative electronic health screening tool with integrated personalized feedback about risk behaviors. The CheckED Yourself App (eHA-IPF) will be divided into an assessment about risk behaviors and a personalized feedback portion. Participants will be randomized to a control or intervention group at the time of consent. Those in the intervention group will receive both parts of the CheckED Yourself App, while the control group will receive only the assessment with no feedback.

Those in the Intervention arm will complete the health risk behavior assessment and receive integrated personalized feedback from the CheckED Yourself App (eHA-IPF), and those in the control group will complete the health risk behavior assessment only. Participants will complete the questionnaire at some point during their ED visit and prior to discharge.

Follow-up assessments will be completed at 1-day and 3 months post ED visit via an online survey. Reminders for the 1-day and 3-month follow-ups will be sent via email or text message. The 1-day assessment will focus on adolescent-reported motivation to make a health behavior change, the content of the ED visit including what, if any, risk behaviors their ED provider discussed with the participant, and satisfaction with care in the ED. The 3-month assessment will include a re-assessment of risk behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 13-18 years of age
* Ability of patient and parent of patient <18 years old to fluently speak and read English
* Has email address and/or cell phone

Exclusion Criteria:

* Inability to independently complete the assessment due to intellectual disability
* Acute cognitive impairment due to injury and/or intoxication
* Administration of IV sedation or pain medications during Emergency Department visit
* Presenting to the Emergency Department due to a psychiatric or mental health complaint
* Emergency Department visit results in hospital admission

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Motivation to change | We anticipate measuring this outcome by September 30, 2018, 6 months after recruitment has closed.
  To evaluate if adolescents who received integrated personalized feedback had higher levels of motivation to change their risk behaviors post-Emergency Department visit compared to adolescents who completed the electronic health assessment only and did not receive personalized feedback
Decreased risk behaviors | We anticipate measuring this outcome by September 30, 2018, 6 months after recruitment has closed.
  To evaluate if adolescents who received integrated personalized feedback reported decreased risk behaviors 3 months post-Emergency Department visit compared to adolescents who completed the electronic health assessment only and did not receive personalized feedback.
Prevalence of risk behaviors | We anticipate measuring this outcome by September 30, 2018, 6 months after recruitment has closed.
  To describe the prevalence of risk behaviors among adolescents who present to the Emergency Department for care.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
N/A IPD will not be shared